CLINICAL TRIAL: NCT02624115
Title: 18F-Fluoroazomycin Arabinoside (FAZA) Positron Emission Tomography/Magnetic Imaging Resonance (PET/MRI) as a Biomarker of Hypoxia in Rectal Cancer: A Pilot Study
Brief Title: FAZA PET as Biomarker for Hypoxia in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 15-9741
Record Dates: First submitted 2015-11-25; First posted 2015-12-08 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Colon Rectal Cancer Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

SUMMARY:
Colorectal cancer (CRC) is one of the leading causes of cancer mortality in Canada. Rectal cancers are now known to be hypoxic which is a negative prognostic factor and predictive of metastatic spread and poor responsiveness to treatment. This has also been shown in preclinical xenograft models. Hence there is a need for identification of hypoxic rectal cancers.

In this pilot study the investigators intend to non-invasively assess the tumor and nodal metastasis using an integrated Positron Emission Tomography-Magnetic Resonance Imaging scanner (PET/MRI) with 18F-Fluoroazomycin Arabinoside (18F-FAZA) a radiopharmaceutical for assessing tumor hypoxia. The hypoxic rectal tumors will show an increased uptake of 18F-FAZA on PET which will have morphological correlation on MRI. The patient will then undergo neoadjuvant chemoradiation therapy (CRT) followed by repeat 18F-FAZA PET/MRI and rectal cancer surgery with pimonidazole staining. Pimonidazole is an extrinsic marker of hypoxia that is selectively reduced and covalently bound to intracellular macromolecules in areas of hypoxia within normal and tumor tissue with current approval for use in humans for research studies.

The primary goal of this pilot trial is to validate FAZA-PET as a biomarker of hypoxia by correlating its uptake in rectal tumors to pimonidazole staining in histopathology specimens. If the investigators pilot study successfully demonstrates the uptake and correlation of pimonidazole and FAZA-PET, the investigators would like to initiate a larger study examining hypoxia in rectal cancer. The investigators aims would be to image patients with locally advanced rectal cancer before CRT to ascertain whether high FAZA-PET uptake correlates with poor outcome to CRT. The ability to preoperatively predict the patient sub-population that will respond best to CRT, will help to identify the "complete pathological" responders and avoid unnecessary surgery. Furthermore, the FAZA-PET high subset of patients may benefit from other treatment strategies including clinical trials of anti-hypoxic agents.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the leading causes of cancer mortality in Canada. Rectal cancers are now known to be hypoxic which is a negative prognostic factor and predictive of metastatic spread and poor responsiveness to treatment. This has also been shown in preclinical xenograft models. Hence there is a need for identification of hypoxic rectal cancers.

In this pilot study, the investigators intend to non-invasively assess the tumor and nodal metastasis using an integrated PET/MRI with a radiopharmaceutical for assessing tumor hypoxia. The hypoxic rectal tumors will show increased uptake of 18F-FAZA on PET which will have morphological correlation on MRI. The patient will then undergo neoadjuvant chemoradiation therapy (CRT) followed by repeat 18F-FAZA PET/MRI and rectal cancer surgery with pimonidazole staining. Pimonidazole is an extrinsic marker of hypoxia that is selectively reduced and covalently bound to intracellular macromolecules in areas of hypoxia within normal and tumor tissue with current approval for use in humans for research studies.

The primary goal of this pilot trial is to validate FAZA-PET as a biomarker of hypoxia by correlating its uptake in rectal tumors to pimonidazole staining in histopathology specimens. If this pilot study successfully demonstrates the uptake and correlation of pimonidazole and FAZA-PET, the investigators would like to initiate a larger study examining hypoxia in rectal cancer. The aim would be to image patients with locally advanced rectal cancer before CRT to ascertain whether high FAZA-PET uptake correlates with poor outcome to CRT. The ability to preoperatively predict the patient subpopulation that will respond best to CRT, will help to identify the "complete pathological" responders and avoid unnecessary surgery. Furthermore, the FAZA-PET high subset of patients may benefit from other treatment strategies including clinical trials of anti-hypoxic agents.

Project Synopsis: STUDY OVERVIEW:

OBJECTIVES:

Primary Objective

1. To determine the feasibility of using the FAZA-PET to image primary tumor hypoxia in patients with rectal cancer prior to treatment with chemoradiotherapy Secondary Objectives
2. To optimize FAZA PET/MRI imaging protocol for use in patients with rectal cancer.
3. To determine whether there is correlation between FAZA-PET, blood oxygen level-dependent MRI and Pimonidazole staining in primary rectal tumors before and after CRT.
4. To correlate hypoxia defined by FAZA PET uptake and blood oxygen level-dependent MRI in rectal cancer with (pathologic) response to neoadjuvant chemoradiotherapy.

Study design: Single arm feasibility pilot study Study scheme: (see below)

Details on Tumor Microscopy and Pimonidazole Image analysis:

The initial assessment of pimonidazole-detected hypoxia in tumor sections from surgical specimens will be immunohistochemical which allows for both qualitative and quantitative assessment of pimonidazole staining in the context of histopathological morphology. To account for heterogeneity of pimonidazole staining, analysis will be performed in multiple surgical sections for each patient tumor (as previously published by the investigators own group). All staining, handling and processing of tissue specimens will done by the pathology department.

STUDY SCHEMA:

Target Population:

* Age ≥ 18 years
* Histological diagnosis of rectal cancer
* Intent to treat with neoadjuvant chemoradiotherapy and surgery
* Negative pregnancy test (for females in child bearing age)

  1. Informed Consent
  2. FAZA-PET/MRI
* Void bladder
* FAZA injection
* Dynamic PET acquisition with MRI Dixon sequences for attenuation correction (60 min; optional )
* 60 minute uptake time (rest)
* Void bladder
* Static PET/MRI pelvis (approximately 45 min)

  3. Standard treatment (neoadjuvant chemoradiotherapy

  4. Oral Pimonidazole on day prior to surgery

  5. Surgery

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion in this study if they meet all of the following criteria:

1. Age ≥18 years
2. Histologic proven locally advanced rectal cancer (T3-T4, or N1) based on clinical assessment and standard staging procedures.
3. Intention to treat with neoadjuvant chemoradiotherapy prior to surgery, according to the current institutional treatment policies.
4. A negative urine or serum pregnancy test within the two week interval immediately prior to imaging, in women of child-bearing age.
5. Ability to provide written informed consent to participate in the study (for both components of the trial: imaging with FAZA-PET/MR and administration of Pimonidazole).

Exclusion Criteria:

Patients will be ineligible to participate in this study if they meet any of the following criteria:

1. Contraindication for MR as per current institutional guidelines.
2. Inability to lie supine for at least 45 minutes.
3. Contraindication for administration of pimonidazole (allergy)
4. Any patient who is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer undergoing neoadjuvant chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-06-09 (Actual); Study Completion 2019-06-09 (Actual)

PRIMARY OUTCOMES:
FAZA PET uptake in locally advanced rectal cancers prior to and after chemoradiotherapy | 1.5 years
  FAZA uptake will be measured by Semiquantitative Uptake Value measurements as well as against a standard of reference (blood pool activity, physiological muscle uptake).

SECONDARY OUTCOMES:
Correlation of FAZA-PET and blood oxygen level-dependent MRI to Pimonidazole staining in locally advanced rectal cancer | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine O'Brien, MD, Principal Investigator — University Health Network, Toronto; Ur Metser, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided